CLINICAL TRIAL: NCT02112006
Title: A Comparison Of Distal Peripheral Nerve Blockade Versus Traditional Proximal Approaches For Hand Surgery
Brief Title: Comparing Two Injection Sites of Local Anesthetic for Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jose Soberon, MD (Other)
Responsible Party: Sponsor-Investigator, Jose Soberon, MD, Anesthesiologist, Ochsner Health System
Organization: Ochsner Health System (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soberon Forearm
Record Dates: First submitted 2014-04-08; First posted 2014-04-11 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2015-10

CONDITIONS: Hand Injury; Wrist Injury; Finger Injury
Keywords: hand surgery; wrist surgery; finger surgery; anesthesia; regional anesthesia; postoperative pain
MeSH Terms: conditions — Hand Injuries; Wrist Injuries; Finger Injuries; Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- distal injection (Experimental): 0.5% bupivacaine injected in the forearm
  Interventions: Procedure: 0.5% bupivacaine injected in the forearm
- proximal injection (Active Comparator): 20-30ml of 0.5% bupivacaine
  Interventions: Procedure: 20-30ml of 0.5% bupivacaine.

INTERVENTIONS:
Procedure: 0.5% bupivacaine injected in the forearm — Median, Ulnar, and Radial nerve blocks performed in the forearm
  Arms: distal injection
Procedure: 20-30ml of 0.5% bupivacaine. — supraclavicular, infraclavicular, or axillary nerve block using 20-30ml of 0.5% bupivacaine.
  Arms: proximal injection

SUMMARY:
The purpose of this study is to compare two different injection sites for local anesthesia in patients having hand surgery. The hypothesis is that subjects receiving injections around the three nerves of the forearm will provide faster pain control and greater patient satisfaction than patients having one injection closer to the shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years of age undergoing unilateral hand, wrist, or finger surgery
* Ability to understand and provide informed consent
* American Society of Anesthesiologists (ASA) status I-III

Exclusion Criteria:

* Patient refusal or inability to provide informed consent
* True allergy, not sensitivity, to any of the following substances: Local Anesthetics, Midazolam, Fentanyl, Hydromorphone, Propofol
* Pregnancy
* Severe hepatic impairment
* Evidence of infection at or near the proposed needle insertion site
* Any sensorimotor deficit of the ipsilateral upper extremity, whether acute or chronic, as determined by the PI and designee
* Pulmonary disease of any kind that is uncontrolled or severe in nature
* Chronic pain patients, defined as someone diagnosed with chronic pain or a chronic pain condition, under the care of a chronic pain physician, or taking oral/intravenous narcotics consistently for 30 days prior to surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
success of block | up to 30 minutes after injection
  number of participants that needed additional anesthesia

SECONDARY OUTCOMES:
pain scores | up to 10 days after surgery
  change in pain scores

OTHER OUTCOMES:
time to complete injection | up to 30 minutes
  difference between the end of injection time and the beginning

CONTACTS AND LOCATIONS:
Overall Officials: Jose Soberon, MD, Principal Investigator — Ochsner Health System
Locations (1):
- Ochsner Clinic Foundation, New Orleans, Louisiana, United States